CLINICAL TRIAL: NCT05834062
Title: Phentermine/Topiramate as Preventive Pharmacotherapy for Obesity
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The project was not funded
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEDS-2022-31025
Record Dates: First submitted 2023-04-13; First posted 2023-04-28 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity | interventions — Qsymia

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Medication arm (Experimental): Individuals randomized to this group will be offered lifestyle-based weight gain prevention counseling. Participants will initiate treatment at 3.75 mg/23 mg orally once in the morning for 14 days, which will then be increased to 7.5 mg/46 mg orally once daily in the morning for the remainder of the trial. Participants who are unable to tolerate the dosing regimen will be maintained at the maximally tolerated dose. To further safeguard the risk/benefit balance we will utilize a down-titration protocol for participants who experience a reduction in BMI below a threshold of 20 kg/m2. In this case, participants will be reduced to the lowest-dose level (3.75 mg/23 mg) for 12 weeks. If the BMI remains below 20 kg/m2 at the lowest dose after 12 weeks, active treatment will be fully withdrawn.
  Participants at the end of the study will be down-titrated gradually with instructions to take the medication every other day for 7 days before stopping treatment altogether.
  Interventions: Drug: Qsymia and lifestyle management therapy
- Placebo arm (Placebo Comparator): Individuals randomized to this group will be offered lifestyle-based weight gain prevention counseling. Participants will initiate treatment with a placebo (to keep the blind) and be asked to up-titrate the placebo dose after the first 14 days and then maintain the placebo dose for the remainder of the study.
  Individuals who are unable to tolerate the dosing regimen will have a down-titration protocol (to maintain the blind) as described in the medication arm. Likewise, we will employ a down-titration protocol for participants who experience a reduction in BMI below a threshold of 20 kg/m2. In this case, participants would be reduced to the lowest dose level of placebo for 12 weeks. If the BMI remains below 20 kg/m2 after 12 weeks, placebo treatment will be fully withdrawn.
  Individuals in the placebo arm will also have a placebo-based down-titration with instructions to take the placebo every other day for 7 days before stopping treatment altogether, to maintain the blind.
  Interventions: Behavioral: Placebo and lifestyle management therapy

INTERVENTIONS:
Drug: Qsymia and lifestyle management therapy — Qsymia will be used at 3.7g mg/23 mg for 12 weeks and then increased to 7.5 mg/46 mg for the remainder of the study. Participants will be offered lifestyle management therapy.
  Arms: Medication arm
Behavioral: Placebo and lifestyle management therapy — Placebo will be used in lieu of Qsymia to maintain the blind. Participants will be offered lifestyle management therapy.
  Arms: Placebo arm

SUMMARY:
This study will test the use of phentermine and topiramate compared with placebo in helping adolescents who are at high risk for developing obesity to lose weight

DETAILED DESCRIPTION:
This study will evaluate the effects of preventative pharmacotherapy on body mass index (BMI), as well as incidence of obesity and normal weight, in adolescents at high risk of developing obesity. We hypothesize that 24 months of Qsymia vs. placebo, in combination with lifestyle-based weight gain prevention coaching, will prevent increases in BMI (primary endpoint). More participants in the placebo group will develop obesity (cross the BMI 30 kg/m2 threshold) and more in the Qsymia group will transition to normal weight (drop below a BMI of 25 kg/m2).

All participants, regardless of medication/placebo assignment, will receive the same foundational weight gain prevention coaching throughout the entire study. The weight gain prevention coaching will be delivered individually by master's level behavioral intervention specialists with expertise in nutrition, physical activity, and weight-related behavior change. The multi-phase prevention intervention will start with 6 weekly 30-minute coaching calls followed by monthly 15-minute check-in calls for the remainder of the first year. At the beginning of the second year, a series of 3, 30-minute coaching calls will be held to revisit the information covered in the initial coaching calls, followed by bi-monthly 15-minute check-in calls for the remainder of the second year. The calls will be conducted via videoconference substituted with phone calls if needed.

The weight gain prevention intervention will utilize empirically supported behavior change strategies to help promote healthy dietary intake, physical activity patterns, and modest weight loss and/or prevent weight gain among participants. The intervention is informed by several of our previous weight loss and maintenance trials and the work of others, including weight gain prevention trials in young adult populations. The core prevention intervention is based on a behavioral conceptualization of effective weight management that emphasizes: 1) identifying behaviors in need of change; 2) setting goals for change; 3) monitoring progress; 4) modifying environmental cues to facilitate change; and 5) modifying consequences to motivate change. The intervention will incorporate core behavior change strategies including self-monitoring, stimulus control, modeling, goal setting, and positive reinforcement, which were among the common behavior change elements identified across the 17 treatment arms used in the Early Adult Reduction of weight through LifestYle (EARLY) weight management trials that included the young adult weight gain prevention trials previously referenced.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 to less than 22 years at screening
* BMI >/= 25 to < 30 kg/m^2
* Family history of obesity defined as one biological parent with severe obesity (BMI >/= 35) and/or two biological parents with obesity (BMI >/= 30)
* Age 16 or 17 years old must also have an obesity-related complication/co-morbidity defined as elevated blood pressure (>/= 130 and/or >/= 80 milligrams of mercury [mmHg]) or current use of anti-hypertensive medication, dyslipidemia (triglycerides >/= 150 milligrams/deciliter (mg/dL) and/or HDL cholesterol < 40 mg/dL or current use of cholesterol-lowering medication, diagnosis of obstructive sleep apnea

Exclusion Criteria:

* Tanner stage 1-4
* Diabetes (1 or 2)
* Current or recent (< 6 months prior to enrollment) use of anti-obesity medication(s) and other weight-altering medication(s) (e.g.,, atypical antipsychotics, attention-deficit hyperactivity disorder [ADHD] stimulant)
* Previous bariatric surgery
* Current or recent (< 6 months prior to enrollment) use of medication(s) to treat insulin resistance
* Recent initiation (< 3 months prior to enrollment) of anti-hypertensive or lipid medication(s)
* History of glaucoma
* Current or recent (< 14 days) use of monoamine oxidase inhibitor
* Known hypersensitivity to sympathomimetic amines
* History of treatment with growth hormone
* Patient Health Questionnaire (PHQ) score of >/= 15
* Eating disorder symptoms within 6 months and/r any past medical diagnosis of eating disorder
* Major psychiatric disorder
* Unstable clinically-diagnosed depression
* History of suicide attempt
* Suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last month
* Current pregnancy or breastfeeding
* Plans to become pregnant
* If sexually active, refusal to use 2 forms of birth control
* Tobacco use
* Alanine transaminase (ALT ) or Aspartate transaminase (AST) >/= 2.5 the upper limit of normal
* Bicarbonate < 18 micromoles per liter (mmol/L)
* Creatinine 1.2 mg/dL
* Creatinine clearance of < 50 microliters per minute [mL/min] (Schwartz formula)
* History of seizures
* Uncontrolled hypertension
* History of structural heart defect
* History of clinically significant arrhythmia
* Diagnosed monogenic obesity
* History of cholelithiasis
* History of nephrolithiasis
* Hyperthyroidism
* Untreated thyroid disorder

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-17 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate effects of preventive pharmacotherapy and lifestyle-based weight gain prevention on body mass index between the medication arm and the placebo arm | 24 months
  Change in BMI

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data may be shared with other researchers